CLINICAL TRIAL: NCT00003294
Title: Initial Clinical Evaluation of the Combination of Paclitaxel and Carboplatin With Modulation of Toxicity With GCSF and Amifostine
Brief Title: Chemotherapy Given With Amifostine and Filgrastim in Treating Patients With Recurrent or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066227; P30CA016056 (NIH); RPCI-DS-97-14; NCI-G98-1410
Record Dates: First submitted 1999-11-01; First posted 2004-08-13 (Estimated); Last update posted 2011-03-07 (Estimated); Status verified 2011-03

CONDITIONS: Leukemia; Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; recurrent adult Hodgkin lymphoma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone | interventions — Filgrastim; Amifostine; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: amifostine trihydrate
Drug: carboplatin
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Chemoprotective drugs such as amifostine may protect normal cells from the side effects of chemotherapy. Colony-stimulating factors such as filgrastim may increase the number of immune cells found in bone marrow or peripheral blood and may help a person's immune system recover from the side effects of chemotherapy.

PURPOSE: Phase I trial to study the effectiveness of combination chemotherapy consisting of paclitaxel plus carboplatin given with amifostine and filgrastim in treating patients with recurrent or metastatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Establish the maximum tolerated dose of a paclitaxel and carboplatin combination modulated by amifostine and filgrastim (G-CSF) in patients with recurrent or metastatic cancer. II. Define the dose limiting toxicity of this combination in these patients. III. Observe any antitumor responses in patients treated with this combination.

OUTLINE: This is a dose escalation study of paclitaxel. Patients receive a 10 minute infusion of amifostine followed by paclitaxel given intravenously over 3 hours followed by carboplatin given over 30 minutes. Filgrastim (G-CSF) is given subcutaneously daily for up to 10 days by self administration starting the following day. Treatment repeats every 28 days for at least 3 courses unless disease progression or unacceptable toxicity occurs. Patients who develop dose-limiting toxicity (DLT) on a given course receive one dose level lower on the next and subsequent courses. Patients with stable disease may continue treatment for as long as benefit is shown. In the absence of DLT in the first 3 patients treated, subsequent cohorts of 3 patients each receive escalating doses of paclitaxel on the same schedule. If DLT occurs in 1 of 3 patients at a given dose level, then 3 additional patients are added at that dose. If DLT occurs in 1 additional patient, this dose is the maximum tolerated dose (MTD); if DLT occurs in more than 2 patients, then 3 additional patients are added at the previous dose. If DLT occurs in no more than 2 of 6 patients, this dose is considered the MTD. At any dose, 3 cases of DLT leads to discontinuation of recruitment at that dose.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent or metastatic malignant disease not amenable to curative surgery, radiotherapy, conventional chemotherapy, or investigational therapy of higher priority Priority given to patients with lung cancer or cancers with tumors easily available for biopsy No CNS disease unless stable post radiation

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 1.5 mg/dL Creatinine clearance at least 50 mL/min Cardiovascular: Systolic blood pressure at least 90 mm Hg No severe heart decompensation No clinically significant cardiac arrhythmia on EKG No inability to tolerate bradycardia Other: No active, uncontrolled infection No nonmalignant systemic disease Not pregnant or nursing Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent immune stimulating agents Chemotherapy: At least 3 weeks since chemotherapy (6 weeks since nitrosourea or mitomycin) and recovered No prior paclitaxel or carboplatin No concurrent chemotherapy Endocrine therapy: No concurrent hormone therapy Radiotherapy: At least 3 weeks since radiotherapy to major bone marrow bearing areas and recovered Concurrent radiotherapy allowed for vital indications or pain relief Surgery: At least 3 weeks since surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1997-05; Primary Completion 1999-04 (Actual); Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary N. Schwartz, MD, Study Chair — Norris Cotton Cancer Center
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States